CLINICAL TRIAL: NCT06112405
Title: Evaluation of App-based Management of Children's Asthma Based on Real World Data and Randomized Control Trial
Brief Title: Real World App-based CCAAP Management of Children With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Capital Institute of Pediatrics, China (Other); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Kunling Shen, Professor, Beijing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BeijingChildrens
Record Dates: First submitted 2023-09-18; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: asthma; children; action plan; App-based
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-based CCAAP (Other): Patients in this group will be provided App-based CCAAP to remind them take medicine regularly and direct them what to do when asthma get worse.
  Interventions: Other: App-based CCAAP
- written CCAAP (Other): Patients in this group will be provided written asthma action plan and direct them what to do when asthma get worse.
  Interventions: Other: Written CCAAP

INTERVENTIONS:
Other: App-based CCAAP — App-based CCAAP, could remind patients take controller and reliever when asthma symptoms get worse through mobile.
  Arms: App-based CCAAP
Other: Written CCAAP — Written CCAAP, conventional management for patients with asthma, remind them take controller and reliever when asthma symptoms get worse.
  Arms: written CCAAP

SUMMARY:
This study is a multi-center randomized controlled trial of children with asthma. The objective of the study is to compare the App-based efficacy of China Children Asthma Action Plan (CCAAP) and written CCAAP used in management of children with asthma. The main questions are:1. Is the App-based CCAAP effective/feasible in management of children with asthma? 2. Is the App-based CCAAP better than written CCAAP in management of children with asthma?

DETAILED DESCRIPTION:
The study is a multi-center randomized control study.The enrollment period is 3 months. Patients who is in 6-17 years of age will be randomized recruited into two groups: the App-based asthma action plan group and the written CCAAP group. Patients in App group will receive written CCAAP and mobile phone-based asthma self-management APP (Youran Respiratory) which includes an electronic asthma action plan, peak expiratory flow monitor system and Peak Expiratory Flow Meter. Patients in written CCAAP management group will write down the symptoms and PEF in asthma diary. The data of the number of asthma episodes, the improvement of FEV1 , the number of unscheduled medical visits, the score of children's quality of life, the questionnaire of asthma knowledge, ACT / C-ACT score, the absent days of parental work, the absent days of children study, and the cost of health economics will be collected regularly in a year with the interval of 3 months to assess the efficacy of CCAAP in asthma management. The study will recruit 400 cases for each group from ten children's hospitals. The study will be completed in a year.

ELIGIBILITY:
Inclusion Criteria:

* did not receive control treatment or did not reach well-control;
* can perform spirometry pulmonary function tests;
* parents are skilled in using smartphones and APP apps (Android or IOS);

Exclusion Criteria:

* reach the level of asthma well control;
* can not use the smartphone APP software;
* can not cooperate the test of peak expiratory flow;
* did not treatment coexist respiratory disease effectively (such as sinusitis, obstructive sleep apnea-hypopnea syndrome, etc.);
* combined with other systemic diseases outside the respiratory system (such as leukemia, rheumatoid arthritis, etc.).
* receiving allergen-specific immunotherapy.
* undergoing trial for other medications or instruments.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
number of asthma exacerbation | 12 months
  unscheduled clinics, emergency visiting, hospitalization, absent of school

CONTACTS AND LOCATIONS:
Overall Officials: Maigeng Zhou, Principal Investigator — Center of Diseases Control and Prevention, China

IPD SHARING:
Plan to Share IPD: No